CLINICAL TRIAL: NCT00518440
Title: A Multi-Center Trial to Study Acute Liver Failure in Adults
Acronym: ALFSG
Status: Completed | Type: Observational
Sponsor: William Lee (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, William Lee, Professor, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Other Study IDs: STU 062010-126; 2U01DK058369 (NIH)
Record Dates: First submitted 2007-08-17; First posted 2007-08-20 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Acute Liver Failure; Fulminant Hepatic Failure; Acute Liver Injury
Keywords: Liver disease; Liver injury
MeSH Terms: conditions — Liver Failure, Acute; Liver Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Urine, DNA and Tissue if available are collected and stored at the NIDDK Central Repository
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to collect clinical and epidemiological data as well as serum, plasma, urine, tissue and DNA samples on individuals who have acute liver failure and on individuals who have acute liver injury, a less severe group of patients who have coagulopathy but do not reach the threshold of encephalopathy.

DETAILED DESCRIPTION:
Although ALF is truly an orphan disease affecting only about 2,000 persons per year, its severity, its frequency among young adults, and its high resource utilization justifies the attention paid to it. In addition, ALF has captured the interest and attention of researchers because of its unique pathogenesis and extreme severity, encouraging us to understand the processes underlying all forms of liver injury, by focusing on this most lethal manifestation.

The etiologies associated with ALF have continued to change further over the years with an apparent decline in viral hepatitis, and a remarkable increase in acetaminophen toxicity to its current level of ~44-50% of cases. A further problem in studying ALF is that the number of cases of a specific etiology observed at any one institution are vanishingly small. The earliest goals of the ALF Study then were to more carefully define the etiologies of ALF on a national scale, and to finally allow in-depth study of specific ALF causes such as autoimmune ALF, viral hepatitis and Wilson disease (WD).

A second group of patients worthy of study are those with acute liver injury.It would be of value to study patients destined to possibly have ALF earlier in their illness for several reasons: first, we might be able to better predict who will progress to full liver failure; second, the current definition requiring encephalopathy limits the number of patients available for study at any site; finally, therapeutic trials might have greater efficacy if begun at earlier disease stages.

Patients who are enrolled are referred to ALFSG clinical sites by gastroenterologist/hepatologist and fellows. Detailed clinical data and bio-specimen (sera, urine, plasma, DNA and tissue if available) are collected. Subjects are followed long-term at 6 months and 12 months. Detailed clinical data and sera are collected.

ELIGIBILITY:
ALF Inclusion Criteria:

* Written Informed consent from patient's next of kin
* Altered mentation of any degree (encephalopathy)
* Evidence of moderately severe coagulopathy (INR ≥ 1.5)
* A presumed acute illness onset of less than 26 weeks
* The NIH guidelines on the inclusion of women and minorities as subjects in clinical research will be observed

ALF Exclusion Criteria:

* Cirrhosis patients
* Alcohol induced liver failure
* Known pre-existing chronic liver disease

ALI Inclusion Criteria:

Acetaminophen (APAP) etiology: acute illness < 2 wks

* INR ≥ 2.0, ALT ≥ 10X ULN Non-acetaminophen etiology: acute illness < 26 wks
* INR≥ 2.0, ALT≥ 10X ULN, TBili ≥ 3 mg/dl

ALI Exclusion Criteria:

• Altered mentation of any degree (encephalopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have acute liver injury or acute liver failure and meet inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 3488 (Actual)
Dates: Start 1998-01; Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: William M Lee, MD, Principal Investigator — University of Southwestern Medical Center
Locations (12):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Francisco, San Francisco, California
  - Yale Medical School, New Haven, Connecticut
  - Northwestern University Medical School, Chicago, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington, Seattle, Washington
- University of Alberta, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Vaquero J, Fontana RJ, Larson AM, Bass NM, Davern TJ, Shakil AO, Han S, Harrison ME, Stravitz TR, Munoz S, Brown R, Lee WM, Blei AT. Complications and use of intracranial pressure monitoring in patients with acute liver failure and severe encephalopathy. Liver Transpl. 2005 Dec;11(12):1581-9. doi: 10.1002/lt.20625. PMID 16315300
- [Background] Fontana RJ, Shakil AO, Greenson JK, Boyd I, Lee WM. Acute liver failure due to amoxicillin and amoxicillin/clavulanate. Dig Dis Sci. 2005 Oct;50(10):1785-90. doi: 10.1007/s10620-005-2938-5. PMID 16187174
- [Background] Schiodt FV, Balko J, Schilsky M, Harrison ME, Thornton A, Lee WM; Acute Liver Failure Study Group. Thrombopoietin in acute liver failure. Hepatology. 2003 Mar;37(3):558-61. doi: 10.1053/jhep.2003.50113. PMID 12601353
- [Background] Schiodt FV, Atillasoy E, Shakil AO, Schiff ER, Caldwell C, Kowdley KV, Stribling R, Crippin JS, Flamm S, Somberg KA, Rosen H, McCashland TM, Hay JE, Lee WM. Etiology and outcome for 295 patients with acute liver failure in the United States. Liver Transpl Surg. 1999 Jan;5(1):29-34. doi: 10.1002/lt.500050102. PMID 9873089
- [Background] Metushi IG, Sanders C; Acute Liver Study Group; Lee WM, Uetrecht J. Detection of anti-isoniazid and anti-cytochrome P450 antibodies in patients with isoniazid-induced liver failure. Hepatology. 2014 Mar;59(3):1084-93. doi: 10.1002/hep.26564. Epub 2014 Jan 27. PMID 23775837
- [Background] Karvellas CJ, Cavazos J, Battenhouse H, Durkalski V, Balko J, Sanders C, Lee WM; US Acute Liver Failure Study Group. Effects of antimicrobial prophylaxis and blood stream infections in patients with acute liver failure: a retrospective cohort study. Clin Gastroenterol Hepatol. 2014 Nov;12(11):1942-9.e1. doi: 10.1016/j.cgh.2014.03.011. Epub 2014 Mar 25. PMID 24674942
- [Result] Lee WM. Acetaminophen and the U.S. Acute Liver Failure Study Group: lowering the risks of hepatic failure. Hepatology. 2004 Jul;40(1):6-9. doi: 10.1002/hep.20293. PMID 15239078
- [Result] Vaquero J, Jordano Q, Lee WM, Blei AT; US Acute Liver Failure Study Group. Serum protein S-100b in acute liver failure: Results of the US Acute Liver Failure Study group. Liver Transpl. 2003 Aug;9(8):887-8. doi: 10.1053/jlts.2003.50172. No abstract available. PMID 12884207
- [Result] The acute liver failure study group. Hepatology. 2002 Dec;36(6):1326. doi: 10.1002/hep.510360603. No abstract available. PMID 12447853
- [Result] Murphy EJ, Davern TJ, Shakil AO, Shick L, Masharani U, Chow H, Freise C, Lee WM, Bass NM. Troglitazone-induced fulminant hepatic failure. Acute Liver Failure Study Group. Dig Dis Sci. 2000 Mar;45(3):549-53. doi: 10.1023/a:1005405526283. PMID 10749332
- [Result] Fontana RJ, McCashland TM, Benner KG, Appelman HD, Gunartanam NT, Wisecarver JL, Rabkin JM, Lee WM. Acute liver failure associated with prolonged use of bromfenac leading to liver transplantation. The Acute Liver Failure Study Group. Liver Transpl Surg. 1999 Nov;5(6):480-4. doi: 10.1002/lt.500050607. PMID 10545534
- [Result] Leung PS, Rossaro L, Davis PA, Park O, Tanaka A, Kikuchi K, Miyakawa H, Norman GL, Lee W, Gershwin ME; Acute Liver Failure Study Group. Antimitochondrial antibodies in acute liver failure: implications for primary biliary cirrhosis. Hepatology. 2007 Nov;46(5):1436-42. doi: 10.1002/hep.21828. PMID 17657817
- [Result] Moller HJ, Gronbaek H, Schiodt FV, Holland-Fischer P, Schilsky M, Munoz S, Hassanein T, Lee WM; U.S. Acute Liver Failure Study Group. Soluble CD163 from activated macrophages predicts mortality in acute liver failure. J Hepatol. 2007 Nov;47(5):671-6. doi: 10.1016/j.jhep.2007.05.014. Epub 2007 Jun 21. PMID 17629586
- [Result] Schiodt FV, Ostapowicz G, Murray N, Satyanarana R, Zaman A, Munoz S, Lee WM. Alpha-fetoprotein and prognosis in acute liver failure. Liver Transpl. 2006 Dec;12(12):1776-81. doi: 10.1002/lt.20886. PMID 17133565
- [Result] Rutherford A, Davern T, Hay JE, Murray NG, Hassanein T, Lee WM, Chung RT; Acute Liver Failure Study Group. Influence of high body mass index on outcome in acute liver failure. Clin Gastroenterol Hepatol. 2006 Dec;4(12):1544-9. doi: 10.1016/j.cgh.2006.07.014. Epub 2006 Sep 25. PMID 16996806
- [Result] Lee WM, Brown KE, Young NS, Dawson GJ, Schlauder GG, Gutierrez RA, Fontana R, Rossaro L, Davern T, Lalani E; Acute Liver Failure Study Group. Brief report: no evidence for parvovirus B19 or hepatitis E virus as a cause of acute liver failure. Dig Dis Sci. 2006 Oct;51(10):1712-5. doi: 10.1007/s10620-005-9061-5. PMID 16964546
- [Result] James LP, Alonso EM, Hynan LS, Hinson JA, Davern TJ, Lee WM, Squires RH; Pediatric Acute Liver Failure Study Group. Detection of acetaminophen protein adducts in children with acute liver failure of indeterminate cause. Pediatrics. 2006 Sep;118(3):e676-81. doi: 10.1542/peds.2006-0069. PMID 16950959
- [Result] Davern TJ 2nd, James LP, Hinson JA, Polson J, Larson AM, Fontana RJ, Lalani E, Munoz S, Shakil AO, Lee WM; Acute Liver Failure Study Group. Measurement of serum acetaminophen-protein adducts in patients with acute liver failure. Gastroenterology. 2006 Mar;130(3):687-94. doi: 10.1053/j.gastro.2006.01.033. PMID 16530510
- [Result] Larson AM, Polson J, Fontana RJ, Davern TJ, Lalani E, Hynan LS, Reisch JS, Schiodt FV, Ostapowicz G, Shakil AO, Lee WM; Acute Liver Failure Study Group. Acetaminophen-induced acute liver failure: results of a United States multicenter, prospective study. Hepatology. 2005 Dec;42(6):1364-72. doi: 10.1002/hep.20948. PMID 16317692
- [Result] Schiodt FV, Rossaro L, Stravitz RT, Shakil AO, Chung RT, Lee WM; Acute Liver Failure Study Group. Gc-globulin and prognosis in acute liver failure. Liver Transpl. 2005 Oct;11(10):1223-7. doi: 10.1002/lt.20437. PMID 16184570
- [Result] Wai CT, Fontana RJ, Polson J, Hussain M, Shakil AO, Han SH, Davern TJ, Lee WM, Lok AS; US Acute Liver Failure Study Group. Clinical outcome and virological characteristics of hepatitis B-related acute liver failure in the United States. J Viral Hepat. 2005 Mar;12(2):192-8. doi: 10.1111/j.1365-2893.2005.00581.x. PMID 15720535
- [Result] Lee WM. Acute liver failure in the United States. Semin Liver Dis. 2003 Aug;23(3):217-26. doi: 10.1055/s-2003-42641. PMID 14523675
- [Result] Vaquero J, Polson J, Chung C, Helenowski I, Schiodt FV, Reisch J, Lee WM, Blei AT. Infection and the progression of hepatic encephalopathy in acute liver failure. Gastroenterology. 2003 Sep;125(3):755-64. doi: 10.1016/s0016-5085(03)01051-5. PMID 12949721
- [Result] Schiodt FV, Davern TJ, Shakil AO, McGuire B, Samuel G, Lee WM. Viral hepatitis-related acute liver failure. Am J Gastroenterol. 2003 Feb;98(2):448-53. doi: 10.1111/j.1572-0241.2003.t01-1-07223.x. PMID 12591067
- [Result] Ostapowicz G, Fontana RJ, Schiodt FV, Larson A, Davern TJ, Han SH, McCashland TM, Shakil AO, Hay JE, Hynan L, Crippin JS, Blei AT, Samuel G, Reisch J, Lee WM; U.S. Acute Liver Failure Study Group. Results of a prospective study of acute liver failure at 17 tertiary care centers in the United States. Ann Intern Med. 2002 Dec 17;137(12):947-54. doi: 10.7326/0003-4819-137-12-200212170-00007. PMID 12484709
- [Result] Teo EK, Ostapowicz G, Hussain M, Lee WM, Fontana RJ, Lok AS; US ALF Study Group (Acute Liver Failure). Hepatitis B infection in patients with acute liver failure in the United States. Hepatology. 2001 Apr;33(4):972-6. doi: 10.1053/jhep.2001.23065. PMID 11283862
- [Result] Taylor RM, Davern T, Munoz S, Han SH, McGuire B, Larson AM, Hynan L, Lee WM, Fontana RJ; US Acute Liver Failure Study Group. Fulminant hepatitis A virus infection in the United States: Incidence, prognosis, and outcomes. Hepatology. 2006 Dec;44(6):1589-97. doi: 10.1002/hep.21439. PMID 17133489
- [Result] Parekh NK, Hynan LS, De Lemos J, Lee WM; Acute Liver Failure Study Group. Elevated troponin I levels in acute liver failure: is myocardial injury an integral part of acute liver failure? Hepatology. 2007 Jun;45(6):1489-95. doi: 10.1002/hep.21640. PMID 17538968
- [Result] Schiodt FV, Bangert K, Shakil AO, McCashland T, Murray N, Hay JE, Lee WM; Acute Liver Failure Study Group. Predictive value of actin-free Gc-globulin in acute liver failure. Liver Transpl. 2007 Sep;13(9):1324-9. doi: 10.1002/lt.21236. PMID 17763387
- [Result] Rutherford AE, Hynan LS, Borges CB, Forcione DG, Blackard JT, Lin W, Gorman AR, Shaikh OS, Reuben A, Harrison E, Reddy KR, Le WM, Chung RT; ALF Study Group. Serum apoptosis markers in acute liver failure: a pilot study. Clin Gastroenterol Hepatol. 2007 Dec;5(12):1477-83. doi: 10.1016/j.cgh.2007.08.007. Epub 2007 Oct 29. PMID 17967565
- [Result] Levitsky J, Duddempudi AT, Lakeman FD, Whitley RJ, Luby JP, Lee WM, Fontana RJ, Blei AT, Ison MG; US Acute Liver Failure Study Group. Detection and diagnosis of herpes simplex virus infection in adults with acute liver failure. Liver Transpl. 2008 Oct;14(10):1498-504. doi: 10.1002/lt.21567. PMID 18825709
- [Result] Korman JD, Volenberg I, Balko J, Webster J, Schiodt FV, Squires RH Jr, Fontana RJ, Lee WM, Schilsky ML; Pediatric and Adult Acute Liver Failure Study Groups. Screening for Wilson disease in acute liver failure: a comparison of currently available diagnostic tests. Hepatology. 2008 Oct;48(4):1167-74. doi: 10.1002/hep.22446. PMID 18798336
- [Result] Polson J, Wians FH Jr, Orsulak P, Fuller D, Murray NG, Koff JM, Khan AI, Balko JA, Hynan LS, Lee WM; Acute Liver Failure Study Group. False positive acetaminophen concentrations in patients with liver injury. Clin Chim Acta. 2008 May;391(1-2):24-30. doi: 10.1016/j.cca.2008.01.018. Epub 2008 Jan 26. PMID 18279672
- [Result] Lee WM, Squires RH Jr, Nyberg SL, Doo E, Hoofnagle JH. Acute liver failure: Summary of a workshop. Hepatology. 2008 Apr;47(4):1401-15. doi: 10.1002/hep.22177. PMID 18318440
- [Result] Li J, Zhu X, Liu F, Cai P, Sanders C, Lee WM, Uetrecht J. Cytokine and autoantibody patterns in acute liver failure. J Immunotoxicol. 2010 Jul-Sep;7(3):157-64. doi: 10.3109/15476910903501748. PMID 20039781
- [Result] James LP, Letzig L, Simpson PM, Capparelli E, Roberts DW, Hinson JA, Davern TJ, Lee WM. Pharmacokinetics of acetaminophen-protein adducts in adults with acetaminophen overdose and acute liver failure. Drug Metab Dispos. 2009 Aug;37(8):1779-84. doi: 10.1124/dmd.108.026195. Epub 2009 May 13. PMID 19439490
- [Result] Schiodt FV, Chung RT, Schilsky ML, Hay JE, Christensen E, Lee WM; Acute Liver Failure Study Group. Outcome of acute liver failure in the elderly. Liver Transpl. 2009 Nov;15(11):1481-7. doi: 10.1002/lt.21865. PMID 19877205
- [Result] Forde KA, Reddy KR, Troxel AB, Sanders CM, Lee WM; Acute Liver Failure Study Group. Racial and ethnic differences in presentation, etiology, and outcomes of acute liver failure in the United States. Clin Gastroenterol Hepatol. 2009 Oct;7(10):1121-6. doi: 10.1016/j.cgh.2009.05.029. Epub 2009 Jun 23. PMID 19501192
- [Result] Lee WM, Hynan LS, Rossaro L, Fontana RJ, Stravitz RT, Larson AM, Davern TJ 2nd, Murray NG, McCashland T, Reisch JS, Robuck PR; Acute Liver Failure Study Group. Intravenous N-acetylcysteine improves transplant-free survival in early stage non-acetaminophen acute liver failure. Gastroenterology. 2009 Sep;137(3):856-64, 864.e1. doi: 10.1053/j.gastro.2009.06.006. Epub 2009 Jun 12. PMID 19524577
- [Result] Cote GA, Gottstein JH, Daud A, Blei AT; Acute Liver Failure Study Group. The role of etiology in the hyperamylasemia of acute liver failure. Am J Gastroenterol. 2009 Mar;104(3):592-7. doi: 10.1038/ajg.2008.84. Epub 2009 Feb 17. PMID 19223884
- [Result] Strnad P, Zhou Q, Hanada S, Lazzeroni LC, Zhong BH, So P, Davern TJ, Lee WM; Acute Liver Failure Study Group; Omary MB. Keratin variants predispose to acute liver failure and adverse outcome: race and ethnic associations. Gastroenterology. 2010 Sep;139(3):828-35, 835.e1-3. doi: 10.1053/j.gastro.2010.06.007. Epub 2010 Jun 9. PMID 20538000
- [Result] Reuben A, Koch DG, Lee WM; Acute Liver Failure Study Group. Drug-induced acute liver failure: results of a U.S. multicenter, prospective study. Hepatology. 2010 Dec;52(6):2065-76. doi: 10.1002/hep.23937. Epub 2010 Oct 14. PMID 20949552
- [Result] Gregory B, Larson AM, Reisch J, Lee WM; Acute Liver Failure Study Group. Acetaminophen dose does not predict outcome in acetaminophen-induced acute liver failure. J Investig Med. 2010 Jun;58(5):707-10. doi: 10.231/JIM.0b013e3181db8764. PMID 20305573
- [Result] Stravitz RT, Lefkowitch JH, Fontana RJ, Gershwin ME, Leung PS, Sterling RK, Manns MP, Norman GL, Lee WM; Acute Liver Failure Study Group. Autoimmune acute liver failure: proposed clinical and histological criteria. Hepatology. 2011 Feb;53(2):517-26. doi: 10.1002/hep.24080. Epub 2011 Jan 5. PMID 21274872
- [Result] Khandelwal N, James LP, Sanders C, Larson AM, Lee WM; Acute Liver Failure Study Group. Unrecognized acetaminophen toxicity as a cause of indeterminate acute liver failure. Hepatology. 2011 Feb;53(2):567-76. doi: 10.1002/hep.24060. Epub 2011 Jan 10. PMID 21274877
- [Result] Ajmera V, Xia G, Vaughan G, Forbi JC, Ganova-Raeva LM, Khudyakov Y, Opio CK, Taylor R, Restrepo R, Munoz S, Fontana RJ, Lee WM; Acute Liver Failure Study Group. What factors determine the severity of hepatitis A-related acute liver failure? J Viral Hepat. 2011 Jul;18(7):e167-74. doi: 10.1111/j.1365-2893.2010.01410.x. Epub 2010 Dec 8. PMID 21143345
- [Result] Rutherford A, King LY, Hynan LS, Vedvyas C, Lin W, Lee WM, Chung RT; ALF Study Group. Development of an accurate index for predicting outcomes of patients with acute liver failure. Gastroenterology. 2012 Nov;143(5):1237-1243. doi: 10.1053/j.gastro.2012.07.113. Epub 2012 Aug 8. PMID 22885329
- [Result] Chung RT, Stravitz RT, Fontana RJ, Schiodt FV, Mehal WZ, Reddy KR, Lee WM. Pathogenesis of liver injury in acute liver failure. Gastroenterology. 2012 Sep;143(3):e1-e7. doi: 10.1053/j.gastro.2012.07.011. Epub 2012 Jul 13. No abstract available. PMID 22796239
- [Result] Lee WM, Stravitz RT, Larson AM. Introduction to the revised American Association for the Study of Liver Diseases Position Paper on acute liver failure 2011. Hepatology. 2012 Mar;55(3):965-7. doi: 10.1002/hep.25551. No abstract available. PMID 22213561
- [Result] Dao DY, Seremba E, Ajmera V, Sanders C, Hynan LS, Lee WM; Acute Liver Failure Study Group. Use of nucleoside (tide) analogues in patients with hepatitis B-related acute liver failure. Dig Dis Sci. 2012 May;57(5):1349-57. doi: 10.1007/s10620-011-2013-3. Epub 2011 Dec 25. PMID 22198704
- [Result] Dao DY, Hynan LS, Yuan HJ, Sanders C, Balko J, Attar N, Lok AS, Word RA, Lee WM; Acute Liver Failure Study Group. Two distinct subtypes of hepatitis B virus-related acute liver failure are separable by quantitative serum immunoglobulin M anti-hepatitis B core antibody and hepatitis B virus DNA levels. Hepatology. 2012 Mar;55(3):676-84. doi: 10.1002/hep.24732. Epub 2012 Jan 31. PMID 21987355
- [Result] Taylor RM, Tujios S, Jinjuvadia K, Davern T, Shaikh OS, Han S, Chung RT, Lee WM, Fontana RJ. Short and long-term outcomes in patients with acute liver failure due to ischemic hepatitis. Dig Dis Sci. 2012 Mar;57(3):777-85. doi: 10.1007/s10620-011-1918-1. Epub 2011 Sep 27. PMID 21948394
- [Result] Stravitz RT, Lisman T, Luketic VA, Sterling RK, Puri P, Fuchs M, Ibrahim A, Lee WM, Sanyal AJ. Minimal effects of acute liver injury/acute liver failure on hemostasis as assessed by thromboelastography. J Hepatol. 2012 Jan;56(1):129-36. doi: 10.1016/j.jhep.2011.04.020. Epub 2011 May 19. PMID 21703173
- [Result] Court MH, Freytsis M, Wang X, Peter I, Guillemette C, Hazarika S, Duan SX, Greenblatt DJ, Lee WM; Acute Liver Failure Study Group. The UDP-glucuronosyltransferase (UGT) 1A polymorphism c.2042C>G (rs8330) is associated with increased human liver acetaminophen glucuronidation, increased UGT1A exon 5a/5b splice variant mRNA ratio, and decreased risk of unintentional acetaminophen-induced acute liver failure. J Pharmacol Exp Ther. 2013 May;345(2):297-307. doi: 10.1124/jpet.112.202010. Epub 2013 Feb 13. PMID 23408116
- [Result] Singh S, Hynan LS, Lee WM; Acute Liver Failure Study Group. Improvements in hepatic serological biomarkers are associated with clinical benefit of intravenous N-acetylcysteine in early stage non-acetaminophen acute liver failure. Dig Dis Sci. 2013 May;58(5):1397-402. doi: 10.1007/s10620-012-2512-x. Epub 2013 Jan 17. PMID 23325162
- [Result] Rangnekar AS, Ellerbe C, Durkalski V, McGuire B, Lee WM, Fontana RJ. Quality of life is significantly impaired in long-term survivors of acute liver failure and particularly in acetaminophen-overdose patients. Liver Transpl. 2013 Sep;19(9):991-1000. doi: 10.1002/lt.23688. Epub 2013 Aug 18. PMID 23780824
- [Result] Stravitz RT, Sanyal AJ, Reisch J, Bajaj JS, Mirshahi F, Cheng J, Lee WM; Acute Liver Failure Study Group. Effects of N-acetylcysteine on cytokines in non-acetaminophen acute liver failure: potential mechanism of improvement in transplant-free survival. Liver Int. 2013 Oct;33(9):1324-31. doi: 10.1111/liv.12214. Epub 2013 Jun 19. PMID 23782487
- [Result] Court MH, Peter I, Hazarika S, Vasiadi M, Greenblatt DJ, Lee WM; Acute Liver Failure Study Group. Candidate gene polymorphisms in patients with acetaminophen-induced acute liver failure. Drug Metab Dispos. 2014 Jan;42(1):28-32. doi: 10.1124/dmd.113.053546. Epub 2013 Oct 8. PMID 24104197
- [Result] Karkhanis J, Verna EC, Chang MS, Stravitz RT, Schilsky M, Lee WM, Brown RS Jr; Acute Liver Failure Study Group. Steroid use in acute liver failure. Hepatology. 2014 Feb;59(2):612-21. doi: 10.1002/hep.26678. Epub 2013 Dec 24. PMID 23929808
- [Result] Karvellas CJ, Fix OK, Battenhouse H, Durkalski V, Sanders C, Lee WM; U S Acute Liver Failure Study Group. Outcomes and complications of intracranial pressure monitoring in acute liver failure: a retrospective cohort study. Crit Care Med. 2014 May;42(5):1157-67. doi: 10.1097/CCM.0000000000000144. PMID 24351370
- [Result] Dubin PH, Yuan H, Devine RK, Hynan LS, Jain MK, Lee WM; Acute Liver Failure Study Group. Micro-RNA-122 levels in acute liver failure and chronic hepatitis C. J Med Virol. 2014 Sep;86(9):1507-14. doi: 10.1002/jmv.23987. Epub 2014 Jun 4. PMID 24895202
- [Result] McGill MR, Staggs VS, Sharpe MR, Lee WM, Jaeschke H; Acute Liver Failure Study Group. Serum mitochondrial biomarkers and damage-associated molecular patterns are higher in acetaminophen overdose patients with poor outcome. Hepatology. 2014 Oct;60(4):1336-45. doi: 10.1002/hep.27265. Epub 2014 Aug 25. PMID 24923598
- [Result] Mellinger JL, Rossaro L, Naugler WE, Nadig SN, Appelman H, Lee WM, Fontana RJ. Epstein-Barr virus (EBV) related acute liver failure: a case series from the US Acute Liver Failure Study Group. Dig Dis Sci. 2014 Jul;59(7):1630-7. doi: 10.1007/s10620-014-3029-2. Epub 2014 Jan 25. PMID 24464209
- [Result] Long D, Fix OK, Deng X, Seielstad M, Lauring AS; Acute Liver Failure Study Group. Whole genome sequencing to identify host genetic risk factors for severe outcomes of hepatitis a virus infection. J Med Virol. 2014 Oct;86(10):1661-8. doi: 10.1002/jmv.24007. Epub 2014 Jun 30. PMID 24978929
- [Result] Tujios SR, Hynan LS, Vazquez MA, Larson AM, Seremba E, Sanders CM, Lee WM; Acute Liver Failure Study Group. Risk factors and outcomes of acute kidney injury in patients with acute liver failure. Clin Gastroenterol Hepatol. 2015 Feb;13(2):352-9. doi: 10.1016/j.cgh.2014.07.011. Epub 2014 Jul 11. PMID 25019700
- [Result] Fontana RJ, Ellerbe C, Durkalski VE, Rangnekar A, Reddy RK, Stravitz T, McGuire B, Davern T, Reuben A, Liou I, Fix O, Ganger DR, Chung RT, Schilsky M, Han S, Hynan LS, Sanders C, Lee WM; US Acute Liver Failure Study Group. Two-year outcomes in initial survivors with acute liver failure: results from a prospective, multicentre study. Liver Int. 2015 Feb;35(2):370-80. doi: 10.1111/liv.12632. Epub 2014 Jul 28. PMID 25039930
- [Result] Laursen TL, Sandahl TD, Stoy S, Schiodt FV, Lee WM, Vilstrup H, Thiel S, Gronbaek H; US Acute Liver Failure Study Group. Circulating mannan-binding lectin, M-, L-, H-ficolin and collectin-liver-1 levels in patients with acute liver failure. Liver Int. 2015 Mar;35(3):756-63. doi: 10.1111/liv.12682. Epub 2014 Sep 30. PMID 25203057
- [Result] Woolbright BL, McGill MR, Staggs VS, Winefield RD, Gholami P, Olyaee M, Sharpe MR, Curry SC, Lee WM, Jaeschke H; Acute Liver Failure Study Group. Glycodeoxycholic acid levels as prognostic biomarker in acetaminophen-induced acute liver failure patients. Toxicol Sci. 2014 Dec;142(2):436-44. doi: 10.1093/toxsci/kfu195. Epub 2014 Sep 19. PMID 25239633
- [Result] Rich NE, Sanders C, Hughes RS, Fontana RJ, Stravitz RT, Fix O, Han SH, Naugler WE, Zaman A, Lee WM. Malignant infiltration of the liver presenting as acute liver failure. Clin Gastroenterol Hepatol. 2015 May;13(5):1025-8. doi: 10.1016/j.cgh.2014.09.040. Epub 2014 Sep 30. PMID 25277846
- [Result] Karvellas CJ, Todd Stravitz R, Battenhouse H, Lee WM, Schilsky ML; US Acute Liver Failure Study Group. Therapeutic hypothermia in acute liver failure: a multicenter retrospective cohort analysis. Liver Transpl. 2015 Jan;21(1):4-12. doi: 10.1002/lt.24021. PMID 25308108
- [Result] Speiser JL, Durkalski VL, Lee WM. Random forest classification of etiologies for an orphan disease. Stat Med. 2015 Feb 28;34(5):887-99. doi: 10.1002/sim.6351. Epub 2014 Nov 3. PMID 25366667
- [Result] Foureau DM, Walling TL, Maddukuri V, Anderson W, Culbreath K, Kleiner DE, Ahrens WA, Jacobs C, Watkins PB, Fontana RJ, Chalasani N, Talwalkar J, Lee WM, Stolz A, Serrano J, Bonkovsky HL. Comparative analysis of portal hepatic infiltrating leucocytes in acute drug-induced liver injury, idiopathic autoimmune and viral hepatitis. Clin Exp Immunol. 2015 Apr;180(1):40-51. doi: 10.1111/cei.12558. PMID 25418487
- [Result] Srungaram P, Rule JA, Yuan HJ, Reimold A, Dahl B, Sanders C, Lee WM; Acute Liver Failure Study Group. Plasma osteopontin in acute liver failure. Cytokine. 2015 Jun;73(2):270-6. doi: 10.1016/j.cyto.2015.02.021. Epub 2015 Mar 21. PMID 25802196
- [Result] Basta G, Del Turco S, Navarra T, Lee WM; Acute Liver Failure Study Group. Circulating levels of soluble receptor for advanced glycation end products and ligands of the receptor for advanced glycation end products in patients with acute liver failure. Liver Transpl. 2015 Jun;21(6):847-54. doi: 10.1002/lt.24129. PMID 25825217
- [Result] Speiser JL, Lee WM, Karvellas CJ; US Acute Liver Failure Study Group. Predicting outcome on admission and post-admission for acetaminophen-induced acute liver failure using classification and regression tree models. PLoS One. 2015 Apr 17;10(4):e0122929. doi: 10.1371/journal.pone.0122929. eCollection 2015. PMID 25885260
- [Result] Serper M, Wolf MS, Parikh NA, Tillman H, Lee WM, Ganger DR. Risk Factors, Clinical Presentation, and Outcomes in Overdose With Acetaminophen Alone or With Combination Products: Results From the Acute Liver Failure Study Group. J Clin Gastroenterol. 2016 Jan;50(1):85-91. doi: 10.1097/MCG.0000000000000378. PMID 26166142
- [Result] Rule JA, Hynan LS, Attar N, Sanders C, Korzun WJ, Lee WM; Acute Liver Failure Study Group. Procalcitonin Identifies Cell Injury, Not Bacterial Infection, in Acute Liver Failure. PLoS One. 2015 Sep 22;10(9):e0138566. doi: 10.1371/journal.pone.0138566. eCollection 2015. PMID 26393924
- [Result] Kaur G, Leslie EM, Tillman H, Lee WM, Swanlund DP, Karvellas CJ; US Acute Liver Failure Study Group. Detection of Ophthalmic Acid in Serum from Acetaminophen-Induced Acute Liver Failure Patients Is More Frequent in Non-Survivors. PLoS One. 2015 Sep 25;10(9):e0139299. doi: 10.1371/journal.pone.0139299. eCollection 2015. PMID 26407170
- [Result] Reddy KR, Ellerbe C, Schilsky M, Stravitz RT, Fontana RJ, Durkalski V, Lee WM; Acute Liver Failure Study Group. Determinants of outcome among patients with acute liver failure listed for liver transplantation in the United States. Liver Transpl. 2016 Apr;22(4):505-15. doi: 10.1002/lt.24347. PMID 26421889
- [Result] Stravitz RT, Ellerbe C, Durkalski V, Reuben A, Lisman T, Lee WM; Acute Liver Failure Study Group. Thrombocytopenia Is Associated With Multi-organ System Failure in Patients With Acute Liver Failure. Clin Gastroenterol Hepatol. 2016 Apr;14(4):613-620.e4. doi: 10.1016/j.cgh.2015.09.029. Epub 2015 Dec 10. PMID 26453953
- [Result] Rosen HR, Biggins SW, Niki T, Gralla J, Hillman H, Hirashima M, Schilsky M, Lee WM; Acute Liver Failure Study Group. Association Between Plasma Level of Galectin-9 and Survival of Patients With Drug-Induced Acute Liver Failure. Clin Gastroenterol Hepatol. 2016 Apr;14(4):606-612.e3. doi: 10.1016/j.cgh.2015.09.040. Epub 2015 Oct 20. PMID 26499927
- [Result] Karvellas CJ, Tillman H, Leung AA, Lee WM, Schilsky ML, Hameed B, Stravitz RT, McGuire BM, Fix OK; United States Acute Liver Failure Study Group. Acute liver injury and acute liver failure from mushroom poisoning in North America. Liver Int. 2016 Jul;36(7):1043-50. doi: 10.1111/liv.13080. Epub 2016 Mar 4. PMID 26837055
- [Result] Reuben A, Tillman H, Fontana RJ, Davern T, McGuire B, Stravitz RT, Durkalski V, Larson AM, Liou I, Fix O, Schilsky M, McCashland T, Hay JE, Murray N, Shaikh OS, Ganger D, Zaman A, Han SB, Chung RT, Smith A, Brown R, Crippin J, Harrison ME, Koch D, Munoz S, Reddy KR, Rossaro L, Satyanarayana R, Hassanein T, Hanje AJ, Olson J, Subramanian R, Karvellas C, Hameed B, Sherker AH, Robuck P, Lee WM. Outcomes in Adults With Acute Liver Failure Between 1998 and 2013: An Observational Cohort Study. Ann Intern Med. 2016 Jun 7;164(11):724-32. doi: 10.7326/M15-2211. Epub 2016 Apr 5. PMID 27043883
- [Result] Hillman L, Gottfried M, Whitsett M, Rakela J, Schilsky M, Lee WM, Ganger D. Clinical Features and Outcomes of Complementary and Alternative Medicine Induced Acute Liver Failure and Injury. Am J Gastroenterol. 2016 Jul;111(7):958-65. doi: 10.1038/ajg.2016.114. Epub 2016 Apr 5. PMID 27045922
- [Result] Koch DG, Tillman H, Durkalski V, Lee WM, Reuben A. Development of a Model to Predict Transplant-free Survival of Patients With Acute Liver Failure. Clin Gastroenterol Hepatol. 2016 Aug;14(8):1199-1206.e2. doi: 10.1016/j.cgh.2016.03.046. Epub 2016 Apr 13. PMID 27085756
- [Result] Fontana RJ, Engle RE, Scaglione S, Araya V, Shaikh O, Tillman H, Attar N, Purcell RH, Lee WM; US Acute Liver Failure Study Group. The role of hepatitis E virus infection in adult Americans with acute liver failure. Hepatology. 2016 Dec;64(6):1870-1880. doi: 10.1002/hep.28649. Epub 2016 Jun 23. PMID 27215797
- [Result] Fix OK, Liou I, Karvellas CJ, Ganger DR, Forde KA, Subramanian RM, Boylan A, Hanje J, Stravitz RT, Lee WM; Acute Liver Failure Study Group. Development and Pilot of a Checklist for Management of Acute Liver Failure in the Intensive Care Unit. PLoS One. 2016 May 13;11(5):e0155500. doi: 10.1371/journal.pone.0155500. eCollection 2016. PMID 27176033
- [Derived] Likhitsup A, Su Z, Rule JA, Anouti A, Rao A, Rostami H, Durkalski-Mauldin V, Lee WM, Fontana RJ. The DILI-Inpt Prognostic Score to Identify Hospitalized Idiosyncratic DILI Patients at Risk for Adverse Outcomes. Clin Gastroenterol Hepatol. 2025 Nov 19:S1542-3565(25)00942-5. doi: 10.1016/j.cgh.2025.11.004. Online ahead of print. PMID 41270879
- [Derived] Patel NH, Chen AY, Osiowy C, Durkalski Mauldin V, Lee WM, Coffin CS, Karvellas CJ; US Acute Liver Failure Study Group. Hepatitis B Virus Variants and Cytokine Patterns in Acute Liver Failure and Transplant-Free Survival. Liver Int. 2025 Jul;45(7):e70175. doi: 10.1111/liv.70175. PMID 40540404
- [Derived] Stravitz RT, Fontana RJ, Karvellas C, Durkalski V, McGuire B, Rule JA, Tujios S, Lee WM; Acute Liver Failure Study Group. Future directions in acute liver failure. Hepatology. 2023 Oct 1;78(4):1266-1289. doi: 10.1097/HEP.0000000000000458. Epub 2023 May 16. PMID 37183883
- [Derived] Rao A, Rule JA, Cerro-Chiang G, Stravitz RT, McGuire BM, Lee G, Fontana RJ, Lee WM. Role of Hepatitis C Infection in Acute Liver Injury/Acute Liver Failure in North America. Dig Dis Sci. 2023 Jan;68(1):304-311. doi: 10.1007/s10620-022-07524-6. Epub 2022 May 11. PMID 35546205
- [Derived] Rao A, Rule JA, Hameed B, Ganger D, Fontana RJ, Lee WM. Secular Trends in Severe Idiosyncratic Drug-Induced Liver Injury in North America: An Update From the Acute Liver Failure Study Group Registry. Am J Gastroenterol. 2022 Apr 1;117(4):617-626. doi: 10.14309/ajg.0000000000001655. PMID 35081550
- [Derived] Zechner C, Adams-Huet B, Gregory B, Neyra JA, Rule JA, Li X, Rakela J, Moe OW, Lee WM; Acute Liver Failure Study Group. Hypophosphatemia in acute liver failure of a broad range of etiologies is associated with phosphaturia without kidney damage or phosphatonin elevation. Transl Res. 2021 Dec;238:1-11. doi: 10.1016/j.trsl.2021.07.003. Epub 2021 Jul 21. PMID 34298149
- [Derived] Davis BC, Tillman H, Chung RT, Stravitz RT, Reddy R, Fontana RJ, McGuire B, Davern T, Lee WM; Acute Liver Failure Study Group. Heat stroke leading to acute liver injury & failure: A case series from the Acute Liver Failure Study Group. Liver Int. 2017 Apr;37(4):509-513. doi: 10.1111/liv.13373. Epub 2017 Feb 17. PMID 28128878
- See also: Acute Liver Failure Study Group website — http://www.acuteliverfailure.org

DOCUMENTS (2):
  • Study Protocol (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT00518440/Prot_000.pdf
  • Informed Consent Form (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT00518440/ICF_001.pdf